CLINICAL TRIAL: NCT06584708
Title: Effect of Low-Volume High-Intensity Training vs. Moderate Intensity Continuous Exercise on Rate Pressure Product and Functional Capacity in Individuals With Increased BMI
Brief Title: Effect of Low-Volume HIT vs. MIC Exercise in Individuals With Increased BMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Rec/01817 Asma Rehman
Record Dates: First submitted 2024-09-02; First posted 2024-09-05 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Overweight and Obesity
Keywords: Low volume High intensity training; Moderate Intensity Continous Exercise; Rate Pressure product; Functional capacity; Increased BMI
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-volume High intensity interval training (Experimental): Group A: Low-volume High intensity interval training
  Interventions: Other: Low-volume high intensity interval training
- Moderate intensity continous exercise (Experimental): Group B: Moderate intensity continous exercise
  Interventions: Other: Moderate intensity continuous exercise

INTERVENTIONS:
Other: Low-volume high intensity interval training — Week 1 & 2:
  Warm-up: 10 minutes at 50% THR Work: 1x4 minutes at 80% THR followed by 1*4 minutes Recovery at 50% THR Cool down: 5 minutes at 50% THR Total exercise time: 23 minutes
  Week 3 & 4:
  Warm-up: 10 minutes at 50% THR Work: 2x6 minutes at 80% THR followed by 1*6 minutes Recovery at 50% THR Cool down: 5 minutes at 50% THR Total exercise time: 33 minutes
  Arms: Low-volume High intensity interval training
Other: Moderate intensity continuous exercise — Week 1 & 2:
  Warm-up: 5 minutes at 50% THR Work: 20 minutes at 60% VO 2 THR Cool Down: 5 minutes at 50% THR Total exercise time: 30 minutes
  Week 3 & 4:
  Warm-up: 5 minutes at 50% THR Work: 30 minutes at 60% THR Cool Down: 5 minutes at 50% THR Total exercise time: 40 minutes
  Arms: Moderate intensity continous exercise

SUMMARY:
To compare the effect of low volume high intensity training and moderate intensity continuous exercise on Rate Pressure Product (RPP) and functional capacity. Limited literature available on effectiveness of Low-volume HIIT in comparison of other Aerobic interventions in obese individuals. In our community, people are sedentary and not involved in routine exercise because of increased weight, so Low volume HIIT would be safe and convenient for such individuals to perform. There is also limited studies available on female gender so both genders are included in this study.

DETAILED DESCRIPTION:
Some recent studies suggest that the rising interest for the potential of high- intensity interval training (HIIT) to enhance the metabolic health in overweight adults. HIIT has also been found to induce comparatively fast enhancements in overall-body aerobic capacity and muscle mitochondrial markers in individuals with overweight.

The main advantage of HIIT is that low-volume HIIT protocols can involve a shorter time as compared with MICT, and time limitations have been recognized as a generally reported hurdle to daily exercise involvement.

Latest studies propose that's when compared to moderate intensity continuous training (MICT), HIIT has been shown to produce similar and sometimes better improvements in results such as cardiorespiratory fitness in spite of often demanding a smaller amount of time commitment and lesser energy expenditure. On the other hand, low volume HIIT is still undecided whether this form of physical training is superior, equivalent or inferior to more outdated forms of exercise training such as MICT for the management cardio metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 23-29.9 kg/m 2 (Overweight-Type I Obese)
* Able to do exercise (PAR-Q)

Exclusion Criteria:

* History of chronic diseases and medication use
* Considerable mental or physical disability, neurological or musculoskeletal problems
* Severe personality disorders or drug addiction.
* Pregnant females

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Rate Pressure Product | 2 weeks, 4 weeks
  Changes from baseline to 2 weeks and 4 weeks after the intervention, measured through product of heart rate and systolic blood pressure, is a very reliable indicator of myocardial oxygen demand. An RPP above 20,000 mmHg per minute is considered healthy, whereas anything below 16,000 mmHg is considered insufficient.
Functional Capacity | 2 Weeks, 4 Weeks
  Changes from baseline to 2 weeks and 4 weeks after the intervention, measured through 6 min walk test (6 MWT). It is a submaximal exercise test that can aid in assessing the functional/exercise capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters that an individual covers in 6 min without any support.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Cantonment General Hospital, Saddar, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No